CLINICAL TRIAL: NCT04570631
Title: A Phase 1b, Open-Label Study of Eftozanermin Alfa (ABBV-621) in Combination With Bortezomib and Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Study to Determine Recommended Phase 2 Dose of Intravenous (IV) Eftozanermin Alfa in Combination With IV or Subcutaneous (SC) Bortezomib and Oral Dexamethasone Tablet and to Assess Change in Disease Symptoms in Adult Participants With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20-258; 2020-001983-26 (EudraCT Number)
Record Dates: First submitted 2020-09-23; First posted 2020-09-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma (MM); Relapsed/Refractory Multiple Myeloma; Eftozanermin Alfa; ABBV-621; Bortezomib; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Safety Lead-in (Experimental): Participants will receive escalating doses of eftozanermin alfa in combination with bortezomib and dexamethasone to determine recommended phase 2 dose (RP2D).
  Interventions: Drug: Eftozanermin alfa; Drug: Bortezomib; Drug: Dexamethasone
- Dose Expansion (Experimental): Participants will receive eftozanermin alfa at RP2D determined in Safety Lead-in part in combination with bortezomib and dexamethasone.
  Interventions: Drug: Eftozanermin alfa; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Eftozanermin alfa — Intravenous (IV) infusion
  Other Names: ABBV-621
Drug: Bortezomib — Intravenous (IV) or Subcutaneous (SC) injection
Drug: Dexamethasone — Oral Tablet

SUMMARY:
Multiple myeloma (MM) is a rare cancer caused by abnormal survival of plasma cells (blood cells). Most trial participants with MM relapse (cancer has come back) or become non- responsive to treatment and remission gets shorter after each line of treatment. This is a study to determine recommended Phase 2 dose and change in disease symptoms of eftozanermin alfa in combination with bortezomib and dexamethasone to assess how efficient the treatment is in adult participants with relapsed/refractory (R/R) MM.

Eftozanermin alfa (ABBV-621) is an investigational drug being developed for the treatment of R/R Multiple Myeloma (MM). Study doctors put the participants in 1 of the 2 groups, called treatment arms. Each group receives a different treatment. Participants in one arm will receive different doses of eftozanermin alfa in combination with bortezomib and dexamethasone to determine phase 2 dose (RP2D). Participants in the other arm will receive eftozanermin alfa at RP2D in combination with bortezomib and dexamethasone. Around 40 adult participants with relapsed/refractory multiple myeloma will be enrolled at approximately 20 sites across the world.

Participants will receive eftozanermin alfa as an infusion into the vein in combination with bortezomib as an infusion into the vein or an injection under the skin and oral dexamethasone tablets for 12 cycles. Each cycle is 21 days for cycles 1-8 and 35 days for cycles 9-12.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma (MM) based on standard International Myeloma Working Group (IMWG) criteria.
* Has measurable disease at screening, defined by at least 1 of the following:

  * Serum M-protein >= 1.0 g/dL (>= 10 g/L); OR
  * Urine M-protein >= 200 mg/24 hours; OR
  * Serum free light chain (sFLC) >= 10 mg/dL (100 mg/L), provided serum FLC ratio is abnormal.
* Relapsed or refractory MM after receiving at least 3, but no more than 6 prior lines of therapy, including an immunomodulatory agent (IMiD), proteasome inhibitor (PI), and an anti-CD38 antibody, and has documented disease progression that occurred during or after the most recent therapy.
* Has adequate hematologic, hepatic and renal function as defined in the protocol.
* Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Life expectancy >= 12 weeks.

Exclusion Criteria:

* Received bortezomib as part of the most recent prior therapy.
* Has primary refractory disease defined as disease that is non-responsive.
* Has not achieved a minimal response or better per IMWG criteria with any therapy.
* Has discontinued bortezomib due to toxicity.
* History of chronic liver disease or significant unresolved liver disease; currently active (within the last 6 months) hepatic impairment according to Child-Pugh Classification B or C.
* History of cataract surgery within 6 months prior to study treatment and participant is not anticipated to have cataract surgery during the study treatment period (as assessed by ophthalmological exam at baseline).
* Evidence of (as assessed by ophthalmological exam at baseline) uveitis, neovascular age related macular degeneration, retinal vein or artery occlusion and/or macular edema; no evidence of moderate or worsening diabetic retinopathy, retinal vascular disease or glaucoma (including participants with history of developing increased intraocular pressure after corticosteroid treatment) per clinical discretion of the consulting eye specialist.
* Peripheral neuropathy Grade >= 2 or Grade 1 with pain.
* Receipt of one of the following:

  * Corticosteroids at a dose equivalent to > 4 mg daily of dexamethasone or a single dose of > 40 mg of dexamethasone within 2 weeks prior to first dose.
  * Monoclonal antibodies used for multiple myeloma treatment within 4 weeks prior to first dose of study treatment.
  * Any other systemic therapies used for multiple myeloma treatment within 5 half-lives or 2 weeks prior to first dose, whichever is longer (or 2 weeks if half-life is unknown).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of Eftozanermin Alfa in Combination With Bortezomib and Dexamethasone (Safety Lead-In Arm) | Up to approximately 3 weeks after the first dose of study drug
  RP2D of eftozanermin alfa in combination with bortezomib and dexamethasone will be determined.
Objective Response Rate (ORR) (Dose Expansion Arm) | Up to approximately 44 weeks after the first dose of study drug
  ORR is defined as percentage of participants with a response of partial response (PR) or better per International Myeloma Working Group (IMWG) criteria.

SECONDARY OUTCOMES:
Rate of Very Good Partial Response (VGPR) or Better per IMWG Criteria | Up to approximately 44 weeks after the first dose of study drug
  Percentage of participants with a response of VGPR or better per IMWG criteria will be assessed.
Duration of Response (DOR) for ORR | Up to approximately 44 weeks after the first dose of study drug
  DOR for ORR is defined as the number of days from the date of first response (PR or better) to the date of first occurrence of progressive disease (PD) or death from any cause, whichever occurs first.
Duration of Response (DOR) for VGPR or Better | Up to approximately 44 weeks after the first dose of study drug
  DOR for VGPR or better rate is defined as the number of days from the date of first response (VGPR or better) to the date of first occurrence of PD or death from any cause, whichever occurs first.
Number of Participants With Dose-Limiting Toxicities (DLTs) | Up to approximately 3 weeks after the first dose of study drug
  DLTs are any of the hematologic, nonhematologic toxicities, adverse events (AEs) occurring following administration of study drug as described in the protocol and evaluated by the Investigator and the sponsor.
Number of Participants With Adverse Events (AEs) | Up to approximately 44 weeks after the first dose of study drug
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator will assess the relationship of each event to the use of study drug as being of reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above.
Change in Vital Sign Measurements | Up to approximately 44 weeks after the first dose of study drug
  Change from baseline in vital sign measurements such as systolic and diastolic blood pressure will be assessed.
Electrocardiogram (ECG) | Up to approximately 44 weeks after the first dose of study drug
  Participants with change from baseline in ECG variables will be assessed.
Number of Participants With Abnormal Clinical Laboratory Test Results | Up to approximately 44 weeks after the first dose of study drug
  Number of participants with abnormal clinical laboratory test results like hematology will be assessed.
Trough Concentration (Ctrough) of Eftozanermin Alfa | Up to Day 106
  Serum concentration prior to administration of study drug.
Maximum Serum Concentration (Cmax) of Eftozanermin Alfa | Up to Day 8
  Serum concentration at 15 min after end of infusion.
Antidrug Antibody (ADA)/Neutralizing Antibody (Nab) Assay | Up to approximately 44 weeks after the first dose of study drug
  Serum sample assay for ADA/Nab (Nabs will be analyzed only upon request).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (19):
- United States (5):
  - Duplicate_Emory University, Winship Cancer Institute /ID# 222922, Atlanta, Georgia
  - Norton Healthcare Pavilion /ID# 222918, Louisville, Kentucky
  - Dana-Farber Cancer Institute /ID# 222174, Boston, Massachusetts
  - Duke University Medical Center /ID# 222166, Durham, North Carolina
  - University of Texas Southwestern Medical Center /ID# 223811, Dallas, Texas
- France (5):
  - Institut Paoli-Calmettes /ID# 222307, Marseille, Bouches-du-Rhone
  - CHRU Lille - Hopital Claude Huriez /ID# 222302, Lille, Nord
  - CHU de Nantes, Hotel Dieu -HME /ID# 222303, Nantes, Pays de la Loire Region
  - HCL - Hopital Lyon Sud /ID# 222304, Pierre-Bénite, Rhone
  - Institut Gustave Roussy /ID# 223951, Villejuif, Val-de-Marne
- Germany (4):
  - Duplicate_Universitaetsklinikum Muenster /ID# 222504, Münster, North Rhine-Westphalia
  - Duplicate_Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz /ID# 222372, Mainz, Rhineland-Palatinate
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 223014, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 222258, Hamburg
- Italy (2):
  - Duplicate_Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita /ID# 223224, Rome, Lazio
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST - IRCCS /ID# 223839, Meldola, Reggio Emilia
- Japan (2):
  - Nagoya City University Hospital /ID# 222408, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 239436, Kashiwa-shi, Chiba
- Hospital Duran i Reynals /ID# 222329, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No